CLINICAL TRIAL: NCT02087670
Title: Natriuretic Brain Pro-peptid (Pro-BNP)Changes in Patients With Chronic Heart Failure Enroled in a Controlled, Supervised Exercise Protocol Within a Cardiac Rehabilitation Program
Brief Title: Natriuretic Brain Pro-peptid Changes in Patients With Chronic Heart Failure Within a Cardiac Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Rehabilitacion en Salud (Network)
Collaborators: Clinica Las Americas (Other)
Responsible Party: Principal Investigator, Jesus Alberto Plata Contreras, M.D Epidemiologist, Grupo Rehabilitacion en Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrupoRS0002
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; cardiac rehabilitation; exercise; Natriuretic Brain Pro-peptid
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- controlled, supervised exercise protocol (Active Comparator): controlled, supervised exercise protocol within a cardiac rehabilitation program
  Interventions: Other: controlled, supervised exercise protocol
- community based exercise (Placebo Comparator): educational program and not supervises exercise program
  Interventions: Other: exercise protocol no supervised

INTERVENTIONS:
Other: controlled, supervised exercise protocol — exercise program within a cardiac rehabilitation program
  Arms: controlled, supervised exercise protocol
Other: exercise protocol no supervised — Exercise program at the community
  Arms: community based exercise

SUMMARY:
Evaluate pro-BNP levels, oxygen consumption, functional class, and quality of life in patients with chronic heart failure after participating in an exercise program and compare them baseline and 2 months, with another group who underwent an educational program.

DETAILED DESCRIPTION:
Clinical controlled trial with a double blinded with a aleatory number sequence as the randomization method, patients will be assigned to one of two groups, intervention program (supervises exercise program) and control group (community based exercise)

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, diagnosed with heart failure (NYHA) II-IV for more than six months

Exclusion Criteria:

* patients with NYHA functional class I, who had attended a cardiac rehabilitation program previously, patients with decompensated diabetes mellitus, hypertension difficult to control, ischemic heart disease in the last month, prior pulmonary embolism, chronic obstructive pulmonary disease, restrictive lung disease , aortic stenosis, new episode of atrial fibrillation and musculoskeletal diseases that limit the performance of physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Alberto Plata Contreras, physiatrist, Principal Investigator — Rehabilitation in health research group. Universidad de Antioquia; Ana Milena García Montoya, Resident, Study Chair — Universidad de Antioquia,Rehabilitation in health research group; Sigifredo Ospina, Doctor, Principal Investigator — Hospital Universitario San Vicente Fundación; Luz Helena Lugo Agudelo, physiatrist, Principal Investigator — Universidad de Antioquia, Rehabilitation in health research group
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient with heart failure were recruited since March 2005 to January 2008.
Period: Overall Study
Arm/Group | Controlled, Supervised Exercise Protocol | Community Based Exercise
Started | 20 | 22
Completed | 17 | 20
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controlled, Supervised Exercise Protocol | Community Based Exercise | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 55 (13) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  Colombia | 20 | 22 | 42
Natriuretic Brain pro-peptide [Median (Full Range); unit: pg/ml] | 429 [74 to 2128] | 278 [49 to 2506] | 386 [49 to 2506]
Oxygen Consumption [Mean (Standard Deviation); unit: ml/min] | 832 (228) | 811 (229) | 821 (226)

OUTCOME MEASURES:

1. Primary Outcome: Natriuretic Brain Pro-peptid
Time Frame: 8 weeks
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Controlled, Supervised Exercise Protocol | Community Based Exercise
Number analyzed (Participants) | 19 | 22
pg/ml | 312 [24 to 2312] | 200 [14 to 3481]

2. Secondary Outcome: Oxygen Consumption
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Controlled, Supervised Exercise Protocol | Community Based Exercise
Number analyzed (Participants) | 17 | 20
ml/min | 831 (250) | 919 (298)

ADVERSE EVENTS:
Time Frame: from March 2005 to January 2008 (2 years and 10 months)
Arm/Group | Controlled, Supervised Exercise Protocol | Community Based Exercise
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes